CLINICAL TRIAL: NCT04881474
Title: The Effects Of Intravenous Ibuprofen on Pain, Oxidative Stress and Inflammation With the Assessment of Thiol-Disulfide Homeostasis and C-Reactive Protein Levels in Laparoscopic Hysterectomy Operations
Brief Title: The Effects Of Intravenous Ibuprofen on Pain, Oxidative Stress and Inflammation in Laparoscopic Hysterectomy Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ersin Kahraman, Resident, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LutfiKirdarTRH
Record Dates: First submitted 2021-02-20; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Analgesia; Ibuprofen; Acetaminophen; Oxidative Stress
MeSH Terms: conditions — Agnosia | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ibuprofen and paracetamol (Active Comparator)
  Interventions: Drug: Ibuprofen 800 mg
- paracetamol only (Active Comparator)
  Interventions: Drug: Ibuprofen 800 mg

INTERVENTIONS:
Drug: Ibuprofen 800 mg — 30-minute lasting iv infusion of 800 mg ibuprofen diluted with 0,9% saline via intravenous route every 6 hours.

SUMMARY:
Objective: The aim of this study is to evaluate whether the exposure of oxidative stres in the peroperative period and the postoperative 24th hour can be decreased with the thiol-disulfide homeostasis (TDH) method and C-Reactive Protein (CRP) with intravenous ibuprofen used for postoperative analgesia in patients undergoing total laparoscopic hysterectomy Material and Method: Sixty-nine patients with American Society of Anesthesiologists (ASA) scores I and II who scheduled for laparoscopic hysterectomy were included in the study. The patients were randomly divided into two groups as ibuprofen and paracetamol (Group IP) and paracetamol (Group P) with the sealed envelope method. When the vascular access was established from all patients (T0), after blood was drawn for TDH and CRP measurements, while 30-minute lasting iv infusion of 800 mg ibuprofen diluted with 0,9% isotonic and iv infusion of 1 g paracetamol was started simultaneously, only 1g of paracetamol infusion was administered in Group P. In the IP group 800 mg ibuprofen and 1 g paracetamol, in the P group only paracetamol, the medicines specified for each group administered intravenously every 6 hours. The postoperative pain level in the patients was evaluated at the 1st, 2nd, 6th, 12th and 24th hours with the Visual Analogue Scale (VAS). Rescue analgesia with 1mg/kg tramadol as an iv bolus was applied to patients whose VAS score was 4 and above. Other blood samples for CRP and TDH were taken before insufflation (T1), after desufflation (T2) and at the postoperative 24th hour (T3). Demographic and hemodynamic data of the patients, duration of anesthesia and Trendelenburg position, need for additional analgesia, presence of nausea and vomiting, VAS scores, pathology results, CRP and TDH levels were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Elective Total Laparoscopic Hysterectomy, Aged between 30 and 65, Body Mass Index (BMI) below 35, ASA class I and II

Exclusion Criteria:

* trauma patients to be operated in emergent conditions, ASA risk classification III-IV and more, have a postoperative intensive care indication, Active and clinical symptoms of anemia, Platelet level lower than 30000 / mm3, History of gastrointestinal bleeding in the last 6 months, History of bleeding diathesis or increased Patients at risk of intracerebral hemorrhage, Oliguric and / or need dialysis in the last 1 month before surgery, or have received dialysis, Patients who used a combination of Warfarin, Lithium, Angiotensin Converting Enzyme (ACE) inhibitor and Furosemide medication or who needed to use any analgesic, muscle relaxant or sedative medication within the last 24 hours.

Patients who had a hypersensitivity reaction to any anesthetic or analgesic drug to be used in the study Patients did not want to participate in the study

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Change of native thiol concentration from baseline (preoperative-T0) to each timepoints (T1-T2-T3) | preoperative (T0), 5 minutes before abdominal insufflation (T1), 15 minutes after abdominal desufflation (T2), postoperative 24 th hour (T3)
  oxidative stress determination with native thiol values
Change of total thiol concentration from baseline (preoperative-T0) to each timepoints (T1-T2-T3) | preoperative (T0), 5 minutes before abdominal insufflation (T1), 15 minutes after abdominal desufflation (T2), postoperative 24 th hour (T3)
  oxidative stress determination with total thiol values
Change of disulfide concentration from baseline (preoperative-T0) to each timepoints (T1-T2-T3) | preoperative (T0), 5 minutes before abdominal insufflation (T1), 15 minutes after abdominal desufflation (T2), postoperative 24 th hour (T3)
  oxidative stress determination with disulfide values
Change of disulfide to native thiol ratio from baseline (preoperative-T0) to each timepoints (T1-T2-T3) | preoperative (T0), 5 minutes before abdominal insufflation (T1), 15 minutes after abdominal desufflation (T2), postoperative 24 th hour (T3)
  oxidative stress determination with disulfide to native thiol ratio

SECONDARY OUTCOMES:
Change of C-Reactive Protein concentration from baseline (preoperative-T0) to each timepoints (T1-T2-T3) | preoperative (T0), 5 minutes before abdominal insufflation (T1), 15 minutes after abdominal desufflation (T2), postoperative 24 th hour (T3)
  Determination of the change of inflammatory response with C-Reactive Protein levels.
Comparing of the pain levels between groups (Group P and Group IP) for each timepoints. | postoperative 1st, 2nd, 6th 12th, 24th hours
  Pain level measured by Visual Analogue Scale
Number of patients who needed tramadol for rescue analgesic | From end of the operation to postoperative 24th hours.
  Determination of patient number who needs rescue analgesic (tramadol).
Average consumption of tramadol for each patient who needed rescue analgesic. | From end of the operation to postoperative 24th hours.
  Determination of average tramadol dose as milligrams

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr. Lütfi Kırdar Training and Research Hospital, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 31.12.2021